CLINICAL TRIAL: NCT06783920
Title: EFFECT of MUSIC in Reducing Pain and Anxiety During Copper T380A Intrauterine Device Insertion in Nulliparous Women.
Brief Title: MUSIC Prior to a T380A Intrauterine Device Insertion in Nulliparous Women.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: music IUD
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Intrauterine Device
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music group (Experimental)
  Interventions: Procedure: music
- no-music group (Placebo Comparator)
  Interventions: Procedure: no music

INTERVENTIONS:
Procedure: music — music will be played during the copper IUD insertion
  Arms: music group
Procedure: no music — IUD insertion will be done as usual without music
  Arms: no-music group

SUMMARY:
The aim is to evaluate the role of music in reducing pain and anxiety during copper IUD insertion in nulliparous women

DETAILED DESCRIPTION:
The aim is to evaluate the role of music in reducing pain and anxiety during copper IUD insertion in nulliparous women

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women aged over 18 years of age requesting a copper IUD for contraception who had a negative pregnancy test.

Exclusion Criteria:

* a prior pregnancy greater than 20 weeks of duration

  * currently pregnant or were pregnant within 6 weeks of study entry
  * had a prior attempted or successful IUD insertion
  * had a history of a cervical procedure such as cone biopsy, Loop electrosurgical excision procedure, or cryotherapy any World Health Organization Medical Eligibility Criteria category 3 or 4 precaution to an IUD active vaginitis or cervicitis
  * undiagnosed abnormal uterine bleeding
  * pelvic inﬂammatory disease within the last 3 months
  * ﬁbroids or other uterine abnormalities distorting the uterine cavity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-22 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
pain during IUD insertion | 5 minutes
  pain will be measured by the 10 cm visual analog scale where 0 denotes no pain, and 10 denotes worst pain felt

SECONDARY OUTCOMES:
anxiety during IUD insertion | 5 minutes
  anxiety will be measured by the 10 cm like visual analog scale where 0 denotes no anxiety, and 10 denotes maximal anxiety